CLINICAL TRIAL: NCT02543177
Title: Optimised Procedure in Patients With an Acute Non-ST-segment Elevation Myocardial Infarction and Acute or Chronic Kidney Disease
Brief Title: Optimised Procedure in Patients With NSTEMI and CKD
Acronym: NSTEMI-CKD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough patients recruited
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-088
Record Dates: First submitted 2015-09-04; First posted 2015-09-07 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Non-ST-segment Elevation Myocardial Infarction; Chronic Kidney Disease
Keywords: NSTEMI, CKD
MeSH Terms: conditions — Renal Insufficiency, Chronic; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- group A (Experimental): direct coronary angiography
  Interventions: Procedure: coronary angiography
- group B (Experimental): direct coronary angiography plus ischemic precondition
  Interventions: Procedure: coronary angiography; Procedure: ischemic precondition
- group C (Experimental): delayed coronary angiography; the kidneys will be irrigated prior to coronary angiography
  Interventions: Procedure: coronary angiography; Procedure: prior kidney irrigation
- group D (Experimental): delayed coronary angiography plus ischemic precondition; the kidneys will be irrigated prior to coronary angiography
  Interventions: Procedure: coronary angiography; Procedure: ischemic precondition; Procedure: prior kidney irrigation

INTERVENTIONS:
Procedure: coronary angiography
Procedure: ischemic precondition — four cycles of congestion and flow of blood in the arm of the patient for 5 minutes
  Arms: group B; group D
Procedure: prior kidney irrigation
  Arms: group C; group D

SUMMARY:
Aim of the study is the determination of the ideal timepoint for the treatment of patients with acute Non-ST-segment Elevation Myocardial Infarction (NSTEMI) and an acute or chronic kidney disease (CKD) with a GRACE score < 140. It should be determine if a prompt coronary angiography or the protection of the kidneys from the used contrast agent is more important for the outcome of the patients. Additionally it will be investigated if the ischemic precondition can help to prevent heart damages.

DETAILED DESCRIPTION:
According to international guidelines a coronary angiography has to be performed within 72h for patients with (NSTEMI).

Patients with a GRACE score > 140 belong to the high risk group and the coronary angiography has to be performed within 24h.

Until today for patients with a GRACE score > 140 and an acute or chronic kidney disease (CKD) the best approach is not known even though up to 40% of all NESTMI patients belong to this population. CKD in connection with an NSTEMI is one predictor for short and long term mortality and serious bleeding as a complication of coronary angiography. Additionally patient with CKD are at risk to experience a contrast agent induced aggravation of the CKD right up to a kidney failure. The pre- and post treatment of the kidneys seem to reduce this risk. The irrigation of the kidneys up to 48h prior coronary angiography optimises the kidney function and buffers the aggravation of kidney function caused by fluid loss or abstention at home.

Additionally the influence of ischemic precondition on one arm of the patient will be evaluated in this setting. First studies give a hint that the kidneys may be protected against the contrast agent of the following catheter examination by ischemic precondition.

ELIGIBILITY:
Inclusion Criteria:

* patient with an acute NSTEMI
* patient with a GRACE score < 140
* patient with an acute or a chronic kidney disease (stage 1 - 5)
* patient who agree with the randomized assignment to one of the study groups in written
* signed Informed content prior to study inclusion
* patient who are legally competent at the time of study inclusion

Exclusion Criteria:

* pregnancy
* nursing women
* patient has been committed to an institution by legal or regulatory order
* Mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study
* participation in a parallel clinical trial
* subjects who are in any state of dependency to the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-09; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of coronary adverse events between the four groups | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Michael Becker, Prof., Principal Investigator — Clinic for Cardiology, Pneumology, Angiology and Internal Intensive Medicine (Medical Clinic I)
Locations (1):
- Prof. Dr. Michael Becker, Aachen, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Goldenberg I, Subirana I, Boyko V, Vila J, Elosua R, Permanyer-Miralda G, Ferreira-Gonzalez I, Benderly M, Guetta V, Behar S, Marrugat J. Relation between renal function and outcomes in patients with non-ST-segment elevation acute coronary syndrome: real-world data from the European Public Health Outcome Research and Indicators Collection Project. Arch Intern Med. 2010 May 24;170(10):888-95. doi: 10.1001/archinternmed.2010.95. PMID 20498417
- [Background] Hasdai D, Behar S, Wallentin L, Danchin N, Gitt AK, Boersma E, Fioretti PM, Simoons ML, Battler A. A prospective survey of the characteristics, treatments and outcomes of patients with acute coronary syndromes in Europe and the Mediterranean basin; the Euro Heart Survey of Acute Coronary Syndromes (Euro Heart Survey ACS). Eur Heart J. 2002 Aug;23(15):1190-201. doi: 10.1053/euhj.2002.3193. PMID 12127921
- [Background] Brar SS, Aharonian V, Mansukhani P, Moore N, Shen AY, Jorgensen M, Dua A, Short L, Kane K. Haemodynamic-guided fluid administration for the prevention of contrast-induced acute kidney injury: the POSEIDON randomised controlled trial. Lancet. 2014 May 24;383(9931):1814-23. doi: 10.1016/S0140-6736(14)60689-9. PMID 24856027
- [Background] Hamm CW, Bassand JP, Agewall S, Bax J, Boersma E, Bueno H, Caso P, Dudek D, Gielen S, Huber K, Ohman M, Petrie MC, Sonntag F, Uva MS, Storey RF, Wijns W, Zahger D; ESC Committee for Practice Guidelines. ESC Guidelines for the management of acute coronary syndromes in patients presenting without persistent ST-segment elevation: The Task Force for the management of acute coronary syndromes (ACS) in patients presenting without persistent ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2011 Dec;32(23):2999-3054. doi: 10.1093/eurheartj/ehr236. Epub 2011 Aug 26. No abstract available. PMID 21873419
- [Background] Szummer K, Lundman P, Jacobson SH, Schon S, Lindback J, Stenestrand U, Wallentin L, Jernberg T; SWEDEHEART. Relation between renal function, presentation, use of therapies and in-hospital complications in acute coronary syndrome: data from the SWEDEHEART register. J Intern Med. 2010 Jul;268(1):40-9. doi: 10.1111/j.1365-2796.2009.02204.x. Epub 2009 Dec 3. PMID 20210836
- [Background] Er F, Nia AM, Dopp H, Hellmich M, Dahlem KM, Caglayan E, Kubacki T, Benzing T, Erdmann E, Burst V, Gassanov N. Ischemic preconditioning for prevention of contrast medium-induced nephropathy: randomized pilot RenPro Trial (Renal Protection Trial). Circulation. 2012 Jul 17;126(3):296-303. doi: 10.1161/CIRCULATIONAHA.112.096370. Epub 2012 Jun 26. PMID 22735306
- [Background] Bae EH, Lim SY, Cho KH, Choi JS, Kim CS, Park JW, Ma SK, Jeong MH, Kim SW. GFR and cardiovascular outcomes after acute myocardial infarction: results from the Korea Acute Myocardial Infarction Registry. Am J Kidney Dis. 2012 Jun;59(6):795-802. doi: 10.1053/j.ajkd.2012.01.016. Epub 2012 Mar 23. PMID 22445708